CLINICAL TRIAL: NCT05503537
Title: Effect of Post-isometric Relaxation Technique and Static Stretching on Length of the Calf Muscles in Post-CABG Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/13
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Bypass
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This study is randomized controlled trial which consist of three group. One group will be given generalized cardiac rehabilitation protocol. Second group will be given post-isometric relaxation technique along with generalized cardiac protocol and third group will be given static stretching along with generalized cardiac protocol. All the groups will be recruited concurrently.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor does not know that the participant receives which treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basic Cardiac Rehabilitation protocol (Active Comparator): ankle pumps and leg slides, 2 sets of 10 repetitions of each exercise. Walk for 10 minutes.
  Interventions: Procedure: Basic Cardiac Rehabilitation Protocol
- post-isometric relaxation technique with basic cardiac protocol (Experimental): ankle pumps and leg slides, 2 sets of 10 repetitions of each exercise. Walk for 10 minutes. Post-isometric relaxation technique: contraction time 10 second using 20% of strength with 15 second rest period in between contractions + 4 repetitions.
  Interventions: Procedure: post-isometric relaxation technique; Procedure: Basic Cardiac Rehabilitation Protocol
- static stretching with basic cardiac protocol (Experimental): Ankle pumps and leg slides, 2 sets of 10 repetitions of each exercise. Walk for 10 minutes. Static stretching: 5 repetitions with 15 sec hold time of stretch.
  Interventions: Procedure: Static stretching; Procedure: Basic Cardiac Rehabilitation Protocol

INTERVENTIONS:
Procedure: post-isometric relaxation technique — Post-isometric relaxation technique will be performed by asking the patient to contract his calf muscles using 20% of his strength. Maintain the contraction for 10 second with 15 second of rest time between each contractions. A total of 4 contractions will be performed.
  Arms: post-isometric relaxation technique with basic cardiac protocol
Procedure: Static stretching — Static stretching will be performed by asking patient to perform dorsiflexion till the point of discomfort. The patient will hold the stretch for 15 second and 5 repetitions will be performed.
  Arms: static stretching with basic cardiac protocol
Procedure: Basic Cardiac Rehabilitation Protocol — Ankle pumps, leg slides, walking

SUMMARY:
Coronary artery bypass grafting (CABG) is one of the common procedure used in coronary artery disease patients which has significant impact on cardiopulmonary and musculoskeletal systems. In the past, phase 1 rehabilitation after procedure focus on cardiopulmonary system. Lower limb rehabilitation is also important part as it influence the cardiac function. Several studies work on post-CABG patients to improve cardiopulmonary fitness but there is less number of data on calf muscles rehabilitation in post-CABG patients. So this study aims to increase the calf muscle extensibility using post-isometric relaxation technique and static stretching.

DETAILED DESCRIPTION:
Coronary artery bypass grafting is one of the common procedure used for coronary artery disease. It has several musculoskeletal and cardiopulmonary complications. Rehabilitation in post-CABG patients accelerates the healing process. In the past, phase 1 includes cardiopulmonary rehabilitation. In the recent years, musculoskeletal rehabilitation is one of the important part after CABG. Muscle energy technique is used to increase muscle extensibility. Different studies show favourable results of static stretching in increasing length of muscles and also of muscle energy technique in increasing length and strength of muscles. There is less evidence on increasing calf muscle flexibility in post-CABG patients. So this study will investigate the technique effective for increasing calf muscle extensibility in post-CABG patients.

This study will be conduced in Armed Forces Institute of Cardiology & National Institute of Heart Diseases(AFIC & NIHD) using non-probability purposive sampling technique. Sample size has been calculated from open epi tool is 135, 45 in each group. Patients are selected according to the inclusion criteria. Patients will be guided about the risks and benefits of the study, voluntary participation and confidentiality of the data. After taking informed consent patients will be randomly assigned to the groups using sealed envelope method. Length of the calf muscles and lower limb tempertaure will be measured before and immediately after the treatment. Post-isometric relaxation technique is given to one group, static stretching to the second group and basic cardiac rehabilitation protocol to the third group.

Group 1(Experimental group): post-isometric relaxation technique using 20% of strength, contraction time of 10 second with 15 second rest period in between+ 4 repetitions. Leg slides and ankle pumps, 2 sets of 10 repetitions. Walk for 10 minutes.

Group 2(Experimental group): static stretching 15 second hold time for stretch + 5 repetitions. Ankle pumps and leg slides: 2 sets of 10 repetitions. Walk for 10 minutes.

Group 3(Control Group): Ankle pumps and leg slides: 2 sets of 10 repetitions. Walk for 10 minutes.

Psot-isometric relaxation technique: This technique will be performed by asking the patient to contract his calf muscles using 20% of the strength. Maintain the contraction for 10 second with 15 second of rest period in between each contraction in which muscle is being lengthened. A total of 4 repetitions will be performed.

Static stretching: This technique will be performed by asking the patient to perform dorsiflexion till the point of discomfort. The patient will maintain the stretch for 15 second and 5 repetitions will be performed.

Length of calf muscles and temperature of lower limb will be measured immediately after the treatment.

ELIGIBILITY:
Inclusion criteria

* Age 35-75 years
* Both males and females
* Post-CABG patients with saphenous vein grafting
* Post-op day 4 with no post-op complications

Exclusion criteria

* Patient with DVT/Pulmonary Embolism, fever, infection at wound site
* Patient with psychosis, osteoporosis, vascular disease
* Hemodynamically unstable patients

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
length of calf muscles | Immediate after treatment
  The length of soleus and gastrocnemius will be measured by using goniometer. The participant will be in supine position with knee extended and knee flexed to 45 degrees for gastrocnemius and soleus muscle respectively. The axis of the goniometer will be placed on lateral malleolus, moving arm parallel to the fifth metatarsal and stationary arm parallel to lower leg. The patient is asked to perform dorsiflexion and the length is measured by recording the angle of the goniometer.

SECONDARY OUTCOMES:
Lower limb temperature | Immediate after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institute of Cardiology and National Institute of Heart Diseases, Rawalpindi, Punjab Province, Pakistan